CLINICAL TRIAL: NCT01515228
Title: Randomized Comparison of Dual Drug-Eluting Cilotax Stent and Everolimus -Eluting Stent Implantation for DE Novo Coronary Artery DisEase in Patients With DIABETES Mellitus
Brief Title: Comparison of Cilotax Stent and Everolimus -Eluting Stent With Diabetes Mellitus (ESSENCE-DM III)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHEOL WHAN LEE, MD, PhD. (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, CHEOL WHAN LEE, MD, PhD., MD, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVRF2011-11
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Coronary Artery Disease
Keywords: requiring drug eluting stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xience Prime stent (Active Comparator): everolimus eluting stent
  Interventions: Device: Cilotax stent
- Cilotax stent (Experimental): paclitaxel with cilostazol dual drug eluting stent
  Interventions: Device: Xience Prime

INTERVENTIONS:
Device: Xience Prime — everolimus-eluting stent implantation
  Other Names: everolimus-eluting stent
  Arms: Cilotax stent
Device: Cilotax stent — paclitaxel with cilostazol dual drug eluting stent implantation
  Other Names: paclitaxel with cilostazol dual drug eluting stent
  Arms: Xience Prime stent

SUMMARY:
The purpose of this study is to examine the safety and effectiveness of coronary stenting with the Cilotax stent compared to the Xience Prime stent in the treatment of diabetic patients.

DETAILED DESCRIPTION:
Prospective, randomized multi-center trial of 300 patients will be enrolled at 7 centers in Korea. Following angiography, diabetic patients with significant diameter stenosis >50% by visual estimation have documented myocardial ischemia or symptoms of angina, and eligible for stenting without any exclusion criteria will be randomized 1:1 to: a) Cilotax stent vs. b) Xience Prime stent. All patients will be followed for at least 1 year. Angiographic follow-up at 9-months is routinely recommended.

ELIGIBILITY:
Inclusion Criteria:

Clinical:

* Diabetic patients with active treatment (oral agent or insulin)
* Patients with angina and documented ischemia or patients with documented silent ischemia
* Patients who are eligible for intracoronary stenting
* Age > 20 years, < 75 years

Angiographic:

* De novo lesion
* Percent diameter stenosis ≥ 50%
* Reference vessel size ≥ 2.5 mm by visual estimation

Exclusion Criteria:

1. History of bleeding diathesis or coagulopathy
2. Pregnant state
3. Known hypersensitivity or contra-indication to contrast agent and heparin
4. Limited life-expectancy (less than 1 year)
5. ST-elevation acute myocardial infraction requiring primary stenting
6. Characteristics of lesion: left main disease, in-stent restenosis, graft vessels
7. Hematological disease (Neutropenia < 3000/mm3), Thrombocytopenia < 100,000/mm3)
8. Hepatic dysfunction, liver enzyme (ALT and AST) elevation ≥ 3times normal
9. Renal dysfunction, creatinine ≥ 2.0mg/dL
10. Contraindication to aspirin, clopidogrel or cilostazol
11. Contraindication to Paclitaxel or everolimus
12. Left ventricular ejection fraction < 30%
13. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period
14. Non-cardiac co-morbid conditions are present with life expectancy < 1 year or that may result in protocol non-compliance (per site investigator's medical judgment for example: oxygen dependent chronic obstructive pulmonary disease, active hepatitis or severe liver function or kidney disease)

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
In-segment late luminal loss | at 9 month angiographic follow-up

SECONDARY OUTCOMES:
All Death | 12 months
Cardiac death | 12 months
Myocardial infarction | 12 months
Target vessel revascularization (ischemia-driven) | 12 months
Target lesion revascularization (ischemia-driven) | 12 months
Stent thrombosis (by ARC definition) | 12 months
Binary restenosis in both in-stent and in-segment | at 9 month angiographic follow-up
Angiographic pattern of restenosis | at 9 month angiographic follow-up
Procedural success | At discharge from the index hospitalization, an expected average of 3 days.
  achievement of a final diameter stenosis of <30% by QCA using any percutaneous method, without the occurrence of death, Q wave MI, or repeat revascularization of the target lesion during the hospital stay
All Death | 1 month
All Death | 4 months
All Death | 9 months
Cardiac death | 1 month
Cardiac death | 4 months
Cardiac death | 9 months
Myocardial infarction | 1 month
Myocardial infarction | 4 months
Myocardial infarction | 9 months
Target vessel revascularization (ischemia-driven) | 1 month
Target vessel revascularization (ischemia-driven) | 4 months
Target vessel revascularization (ischemia-driven) | 9 months
Target lesion revascularization (ischemia-driven) | 1 month
Target lesion revascularization (ischemia-driven) | 4 months
Target lesion revascularization (ischemia-driven) | 9 months
Stent thrombosis (by ARC definition) | 1 month
Stent thrombosis (by ARC definition) | 4 months
Stent thrombosis (by ARC definition) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Cheol-Whan Lee, MD, Principal Investigator — Asan Medical Center
Locations (9):
- South Korea (9):
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Inje University Pusan Paik Hospital, Pusan
  - Asan Medical Center, Seoul
  - Ulsan University Hospital, Ulsan